CLINICAL TRIAL: NCT05861596
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Dysphagia in Individuals With Stroke
Brief Title: Repetitive Transcranial Magnetic Stimulation on Dysphagia in the Stroke Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Lai chien hung, Professor, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N201912080
Record Dates: First submitted 2023-01-19; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Dysphagia; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Conscript 10 individuals, every individual will receive 20 mins of repetitive transcranial magnetic stimulation and 30 min NMES combined with conventional swallowing therapy, 5 times per week, lasting for 2 weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Device: Neuromuscular electrical stimulation combined with conventional swallowing training
- Group B (Sham Comparator): Conscript 10 individuals, every individual will receive sham repetitive transcranial magnetic stimulation and 30 min NMES combined with conventional swallowing therapy, 5 times per week, lasting for 2 weeks.
  Interventions: Device: Neuromuscular electrical stimulation combined with conventional swallowing training

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Participants suffered from acute stroke with dysphagia in single hospital who were determined by CT/MRI and clinical evaluation. The aim of this study is to compare the effects of rTMS, Neuromuscular electrical stimulation (NMES) and conventional swallowing therapy to those of sham rTMS, Neuromuscular electrical stimulation(NMES) and conventional swallowing therapy. One group will receive Neuromuscular electrical stimulation(NMES), to sham One group will receive Neuromuscular electrical stimulation(NMES),traditional swallowing therapy and rTMS therapy five times per week for 2 weeks ; Another group will receive Neuromuscular electrical stimulation(NMES) and traditional swallowing therapy with shame rTMS five times per week for 2 weeks. MEP character, FEES, degrees of dysphagia, FOIS, and SSA were used for evaluated swallowing function before the therapy and after 2 weeks therapy.
  Arms: Group A
Device: Neuromuscular electrical stimulation combined with conventional swallowing training — Participants suffered from acute stroke with dysphagia in single hospital who were determined by CT/MRI and clinical evaluation. The aim of this study is to compare the effects of rTMS, Neuromuscular electrical stimulation (NMES) and conventional swallowing therapy to those of sham rTMS, Neuromuscular electrical stimulation(NMES) and conventional swallowing therapy. One group will receive Neuromuscular electrical stimulation(NMES), to sham One group will receive Neuromuscular electrical stimulation(NMES),traditional swallowing therapy and rTMS therapy five times per week for 2 weeks ; Another group will receive Neuromuscular electrical stimulation(NMES) and traditional swallowing therapy with shame rTMS five times per week for 2 weeks. MEP character, FEES, degrees of dysphagia, FOIS, and SSA were used for evaluated swallowing function before the therapy and after 2 weeks therapy.

SUMMARY:
Participants suffered from acute stroke with dysphagia in single hospital who were determined by CT/MRI and clinical evaluation. Current project will recruit participants and randomize into two groups.One group will receive NMES, traditional swallowing therapy and rTMS therapy five times per week for 2 weeks ; Another group will receive NMES and traditional swallowing therapy with shame rTMS five times per week for 2 weeks. FEES and SSA were used for evaluated swallowing function before the therapy and after 2 weeks therapy.

DETAILED DESCRIPTION:
Participants suffered from acute stroke with dysphagia in single hospital who were determined by CT/MRI and clinical evaluation. The aim of this study is to compare the effects of rTMS, NMES and conventional swallowing therapy to those of sham rTMS, NMES and conventional swallowing therapy. One group will receive NMES, to sham One group will receive NMES,traditional swallowing therapy and rTMS therapy five times per week for 2 weeks ; Another group will receive NMES and traditional swallowing therapy with shame rTMS five times per week for 2 weeks. MEP character, FEES, degrees of dysphagia, FOIS, and SSA were used for evaluated swallowing function before the therapy and after 2 weeks therapy.

ELIGIBILITY:
Inclusion Criteria:

1. stroke
2. Onset time at least for one week，area not be limited.
3. Patient was first time stroke patient without obvious infection condition.
4. Patients with dysphagia in the stroke who were diagnosed by neurologist and CT/MRI in our institute. Patient was clear with adequate motivation and could cooperate the whole therapy and FEES evaluation.

Exclusion Criteria:

1. Lower motor neuron disease, such as autonomic dysreflexia, facial palsy, hyhoid muscle denervation.
2. Mental status unstable, mental retardation, schizophrenia, bipolar disease were be excluded.
3. Metal implantation of head, ventroperotoneal shunt or any seizure history, pacemaker, as well as head and neck cancer.
4. Allergy to specific subjects
5. Cognition impairment
6. Alcohol or drugs abuse
7. Afraid of the noise of rTMS.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Fiberoptic Endoscopic Examination of Swallowing (FEES) at 2 weeks | one day before intervention, 1 day after intervention
  In this study, FEES is executed before and after intervention. The assessment of FEES is as follows.
  Hyodo-score: for predicting aspiration with moderate sensitivity and high specificity.
  This method consists of four parameters; These four parameters are each scored 0-3 on a 4 point scale (0; normal, 1; mildly impaired, 2; moderately impaired, 3; severely impaired). The Hyodo score is expressed as the sum of scores for each of the four parameters, ranging 0- 12. Patients with a score of less than 5 were assessed as having normal swallowing function. Patients with a score of more than 8 had severe swallowing dysfunction and would not be allowed any oral intake.
Change from baseline in The Fiberoptic Endoscopic Dysphagia Severity Scale (FEDSS) at 2 weeks | one day before intervention, 1 day after intervention
  The Fiberoptic Endoscopic Dysphagia Severity Scale (FEDSS):
  Stroke-related dysphagia was divided into a six-point FEDSS with 1 score for the best and 6 scores for the worst.
Change of baseline Standardized Swallowing Assessment (SSA) at 2 weeks | one day before intervention, 1 day after intervention
  In this study, SSA was executed before and after intervention. SSA is a standard of universal screening of all stroke patients within 24 hours of admission. And SSA comprises three sections and was designed to terminate if a problem was encountered. The first section checked whether the patient was physically capable of screening; sections 2 and 3 comprised the main screening test. Volitional cough, saliva control, oral motor dexterity, respiratory compromise and phonation were first evaluated; if no problems were elicited, the ability to swallow water was observed.
Change of baseline Latency of Motor evoked potentials (MEP) at 2 weeks | one day before intervention, 1 day after intervention
  Onset latency of MEP, The latency, however, may provide information about the stress in damaged motor pathways.
Change of baseline Amplitude of Motor evoked potentials (MEP) at 2 weeks | one day before intervention, 1 day after intervention.
  Onset to peak amplitude of Motor evoked potentials (MEP).The amplitude of motor evoked potentials (MEPs) elicited by transcranial magnetic stimulation (TMS) is a common yet highly variable measure of corticospinal excitability.

SECONDARY OUTCOMES:
Change of baseline Degree of dysphagia at 2 weeks | one day before intervention, 1 day after intervention
  Score of degree of dysphagia, score 0 shows normal swallowing, score 1 is able to swallow , some solid food, score 2 is able to swallow semi-liquid food, score 3 is able to swallow liquids only, score 4 exhibits absolute dysphagia.
Change of Functional Oral Intake Scale (FOIS) at 2 weeks | one day before intervention, 1 day after intervention
  Functional Oral Intake Scale
Change of baseline modified water swallowing test at 2 weeks | one day before intervention, 1 day after intervention
  modified water swallowing test

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Lai, MD, PhD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan